CLINICAL TRIAL: NCT05271162
Title: Evaluation of the Effectiveness of Empagliflozin in the Prevention of Cardiotoxicity in Cancer Patients Undergoing Chemotherapy Based on Anthracyclines (EMPACT Study).
Brief Title: Empagliflozin in the Prevention of Cardiotoxicity in Cancer Patients Undergoing Chemotherapy Based on Anthracyclines
Acronym: EMPACT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Anna Borowiec, Principal Investigator, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ABM/03/00012
Record Dates: First submitted 2022-02-20; First posted 2022-03-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cardiotoxicity
Keywords: Cardiotoxicity; Empagliflozin; Anthracyclines
MeSH Terms: conditions — Cardiotoxicity | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Active Comparator): Empagliflozin, 10 mg q.d; p.o
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Placebo 1 tabl q.d; p.o
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Empagliflozin 10 mg q.d; p.o
  Other Names: Jardiance
  Arms: Empagliflozin
Other: Placebo — Placebo 1 tabl q.d; p.o
  Arms: Placebo

SUMMARY:
EMPACT (EMPAgliflozin in prevention of chemotherapy-related CardioToxicity) study is a randomized, multi-center, placebo-controlled, double-blind trial to evaluate efficacy of empagliflozin in prevention of left ventricular (LV) dysfunction in patients receiving high cumulative doses of anthracyclines. Diagnosed with cancer, 220 patients without history of heart failure and LV ejection fraction (EF) ≥ 50%, scheduled for high dose anthracyclines (doxorubicin ≥240 mg/m2 or epirubicin ≥540 mg/m2), will be included in the study. They will be randomized to a 10 mg of empagliflozin once daily or to matching placebo in a 1:1 ratio. The primary objective of the EMPACT study is to assess whether prophylactic SGLT-2 inhibitors may prevent a reduction in LVEF after high doses anthracyclines, as evaluated by serial echocardiography on each visit and cardiovascular magnetic resonance (CMR) performed at randomization and on its completion. The secondary composite endpoint includes: all-cause death, cardiovascular (CV) death, myocardial infarction and ischemic stroke. Additional secondary outcome measures include structural myocardial alterations assessed by CMR, decrease in GLS (global longitudinal strain) in echocardiography and changes in cardiac biomarkers. The study will be carried out in accordance with GCP and monitoring will be outsourced to a subcontractor - CRO. The examination will be insured and will begin as soon as the required approvals are obtained.

DETAILED DESCRIPTION:
Malignant neoplasms are the second most common cause of death in Poland. Cancer mortality decreased by 27% over the past 25 years. Improved survival in cancer patients is related to several factors, such as prevention, early detection and the introduction of new chemotherapy regimens. However, the benefits of administration of anti-cancer drugs are partially limited by their adverse effects on the cardiovascular system, resulting in increased morbidity and mortality from complications of this treatment. The most serious toxic effect of chemotherapy is damage to the heart muscle leading to its failure, often referred to as 'cardiotoxicity'. This serious complication remains an unresolved clinical problem. The use of doxorubicin is associated with the development of congestive heart failure even in 48% of patients at the doxorubicin total dose of 700 mg/m2. The only drug approved for the prophylactic treatment of cardiac complications is dexrazoxane. However, it is only recommended for patients with advanced breast cancer receiving doxorubicin or epirubicin who have previously received a cumulative dose of 300 mg/m2 of doxorubicin or a cumulative epirubicin dose of 540 mg/m2, when further anthracycline therapy is required. Dexrazoxane is an expensive drug and may influence the effectiveness of chemotherapy. Routine prophylaxis of myocardial dysfunction is not currently recommended due to insufficient data from randomized clinical trials. So far, the prophylactic effects of such cardiological drugs as: angiotensin converting enzyme (ACE) inhibitors and angiotensin receptor blockers (ARBs), beta-blockers, statins and ranolazine have been studied. The results of these studies are contradictory. Therefore, at present, only symptomatic patients with decreased left ventricular ejection fraction or elevated levels of cardiac biomarkers are eligible for treatment with heart failure medications. Empagliflozin is an orally administered once-daily, highly selective sodium-glucose cotransporter 2 (SGLT2) inhibitor proven to treat patients with chronic heart failure of different aetiologies, also with preserved left ventricle systolic function. This drug also has additional nephroprotective, anti-inflammatory and metabolic effects. In recent animal studies, the cardioprotective effect of empagliflozin during the use of anthracyclines was demonstrated.

EMPACT (EMPAgliflozin in prevention of chemotherapy-related CardioToxicity) study is a randomized, multi-center, placebo-controlled, double-blind trial to evaluate efficacy of empagliflozin in prevention of left ventricular (LV) dysfunction in patients receiving high cumulative doses of anthracyclines. Diagnosed with cancer, 220 patients without history of heart failure and LV ejection fraction (EF) ≥ 50%, scheduled for high dose anthracyclines (doxorubicin ≥240 mg/m2 or epirubicin ≥540 mg/m2), will be included in the study. They will be randomized to a 10 mg of empagliflozin once daily or to matching placebo in a 1:1 ratio. The primary objective of the EMPACT study is to assess whether prophylactic SGLT-2 inhibitors may prevent a reduction in LVEF after high doses anthracyclines, as evaluated by serial echocardiography on each visit and cardiovascular magnetic resonance (CMR) performed at randomization and on its completion. The secondary composite endpoint includes: all-cause death, cardiovascular (CV) death, myocardial infarction and ischemic stroke. Additional secondary outcome measures include structural myocardial alterations assessed by CMR, decrease in GLS (global longitudinal strain) in echocardiography and changes in cardiac biomarkers. This is the first study of this type in the world, we hope that the results of this project will change the standards of management of oncological patients and contribute to the improvement of their survival and quality of life.

ELIGIBILITY:
The study will include patients with diagnosed cancer, diagnosed and qualified for further systemic treatment at the National Institute of Oncology in Warsaw. Patients must give informed and voluntary consent to participate in the study and meet all the conditions for inclusion in the study

Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.
2. Age ≥18 years at the time of signing the informed consent.
3. Known neoplastic disease prior to the initiation of chemotherapy with a high dose of anthracyclines (doxorubicin ≥ 240 mg / m2 b.w. or epirubicin ≥ 540 mg / m2 b.w.)
4. No history of heart failure (left ventricular ejection fraction ≥ 50% as assessed by echocardiography).
5. Women of child-bearing age must have a negative serum or urine pregnancy test.
6. All males and females must consent to the use of effective contraception throughout the study period and after study medication is discontinued.
7. Sexually active women of childbearing potential must use 2 effective methods of contraception (abstinence, IUD, oral contraceptive or double barrier device) from informed consent and for at least 6 months after study drug discontinuation
8. Sexually active men and their sexual partners must use effective methods of contraception from the moment they sign their informed consent to participate in the study and for at least 3 months after discontinuation of the study drug.

Exclusion Criteria:

1. History of heart failure
2. Left ventricle systolic dysfunction assessed by echocardiography (LVEF <50%)
3. Significant valve disease
4. Previous chemotherapy or radiation to the chest
5. Symptomatic hypotension and / or SBP <100 mmHg at Visit 1 or Visit 2
6. Liver disease, as determined by ALT, AST, or alkaline phosphatase levels above 3 x upper limit of normal (ULN) at visit 1.
7. Renal impairment, defined as eGFR <20 mL / min / 1.73 m2 or dialysis requirement, as determined at Visit 1.
8. History of ketoacidosis
9. Gastrointestinal surgery or gastrointestinal disturbance that could impair drug absorption
10. Presence of any disease with a life expectancy <1 year in the opinion of the investigator.
11. Treatment with any SGLT-2 inhibitor for up to 3 months prior to study enrollment.
12. Pregnancy or breastfeeding
13. Drug or alcohol abuse
14. Suspected non-compliance and irregular use of study drug
15. Inability to perform CMR, e.g. claustrophobia, weight> 120 kg, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with diagnosis of cancer treatment-related cardiac dysfunction (CTRCD) at any time over the 12-month study period | from date of randomization until 12 months
  CTRCD is defined as decrease in LVEF in echocardiography of at least 10% from baseline to a final LVEF of less than 50% and/or a relative decrease of at least 15% in global longitudinal strain (GLS) from baseline.

SECONDARY OUTCOMES:
Rate of episodes of all-cause death, cardiovascular death, myocardial infarction, and stroke | from date of randomization up to 12 months
  medical records
Percentage decrease in left ventricular ejection fraction, GLS (global longitudinal strain) | from date of randomization up to 12 months
  echocardiography
Rate of structural myocardial alterations in CMR | from date of randomization up to 12 months
  cardiovascular magnetic resonance
Changes in the concentration of biomarkers | from date of randomization up to 12 months
  blood samples, Troponina, NTproBNP
The difference in scores in the KCCQ (Kansas City Cardiomyopathy Questionnaire) assessing the quality of life of patients. | from date of randomization up to 12 months
  Kansas City Cardiomyopathy Questionnaire, the minimum and maximum values:0-100, higher scores mean a better outcome.
The proportion of participants with an absolute decline in LVEF of 10% or greater in LVEF from prior to chemotherapy to a final value of less than 53% over the 12-month study period. | from randomization up to 12 months
  echocardiography
HF hospitalization or Need for outpatient intensification of HF therapy | from randomization up to 12 months
  medical records

CONTACTS AND LOCATIONS:
Overall Officials: Anna Borowiec, PhD, Principal Investigator — Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, POLAND
Locations (2):
- Poland (2):
  - Institute of Hematology and Transfusion Medicine, Warsaw
  - National Institute of Oncology, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: In September For 6 years